CLINICAL TRIAL: NCT00630552
Title: A Phase 1b/2 Study to Evaluate the Safety and Efficacy of AMG 655 or AMG 479 in Combination With Gemcitabine as First-Line Therapy for Metastatic Pancreatic Cancer
Brief Title: QUILT-2.019: A Study of AMG 655 or AMG 479 in Combination With Gemcitabine for Treatment of Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NantCell, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 20060323; QUILT-2.019 (Other: NantCell, Inc.)
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Results first posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Adenocarcinoma of the Pancreas; Metastatic Pancreatic Cancer; Pancreatic Cancer
Keywords: AMG 479; Gemcitabine; TR-2; IGF-1R; AMG 655; Pancreatic cancer; Adenocarcinoma of the Pancreas; Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Insulin-Like Growth Factor I, Resistance To | interventions — ganitumab; conatumumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- Phase 1b AMG 655 3mg/kg (Experimental): Subjects were treated with one of 2 dose levels of AMG 655 (3 mg/kg) with gemcitabine.
  Interventions: Drug: AMG 655
- Phase 1b AMG 655 10mg/kg (Experimental): Subjects were treated with one of 2 dose levels of AMG 655 (10 mg/kg) with gemcitabine.
  Interventions: Drug: AMG 655
- Phase 2 AMG 655 (Experimental): Subjects were treated with the dose of AMG 655 (10mg/kg) in combination with gemcitabine. Gemcitabine (1000 mg/m2) was administered by intravenous infusion on days 1, 8 and 15 of each 28 day cycle followed by the AMG 655 infusion on days 1 and 15 after completion of the gemcitabine infusion.
  Interventions: Drug: AMG 655
- Phase 2 AMG 479 (Experimental): Subjects were treated with the dose of AMG 479 (12 mg/kg) in combination with gemcitabine. Gemcitabine (1000 mg/m2) was administered by intravenous infusion on days 1, 8 and 15 of each 28 day cycle followed by the AMG 479 infusion on days 1 and 15 after completion of the gemcitabine infusion.
  Interventions: Drug: AMG 479
- Phase 2 AMG 655-placebo (Placebo Comparator): Subjects were treated with the dose of AMG 655-placebo in combination with gemcitabine. Gemcitabine (1000 mg/m2) was administered by intravenous infusion on days 1, 8 and 15 of each 28 day cycle followed by the AMG 655-placebo infusion on days 1 and 15 after completion of the gemcitabine infusion.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — Inactive dummy of AMG 655.
  Arms: Phase 2 AMG 655-placebo
Drug: AMG 479 — AMG 479 is fully human monoclonal antagonist antibody targeted against insulin-like growth factor receptor type 1 (IGF-1R).
  Arms: Phase 2 AMG 479
Drug: AMG 655 — AMG 655 is a fully human monoclonal agonist antibody directed against TRAIL Receptor 2 (TR-2).
  Arms: Phase 1b AMG 655 10mg/kg; Phase 1b AMG 655 3mg/kg; Phase 2 AMG 655

SUMMARY:
This is a multi-center, 2-part study of AMG 655, AMG 479 or AMG 655-placebo plus gemcitabine as first-line treatment of subjects with metastatic pancreatic cancer. Part 1 is an open-label, dose-escalation phase 1b segment to determine the safety, tolerability and maximum tolerated dose of AMG 655 in combination with gemcitabine. Enrollment into part 1 of the study has been completed. Part 2 is a randomized, placebo-controlled phase 2 segment to estimate the efficacy as assessed by 6 month survival of AMG 655, AMG 479, or AMG 655-placebo in combination with gemcitabine. The phase 2 segment that will commence after dose selection in part 1. In part 2, subjects will be randomized 1:1:1 to AMG 655, AMG 479, or placebo in combination with gemcitabine.

ELIGIBILITY:
Inclusion Criteria:

* Untreated metastatic adenocarcinoma of the pancreas (AJCC Stage IV)
* Subjects with unresectable pancreatic cancer who have had surgery are eligible if fully recovered and greater than 30 days have elapsed since the surgery.

Subjects with a history of pancreatoduodenectomy are eligible provided that there is radiographically documented disease recurrence.

* Men or women ≥ 18 years of age
* Eastern Cooperative Oncology Group (ECOG) score of 0 or 1
* Adequate hematologic, hepatic, renal and coagulation function
* Amylase and lipase ≤ 2.0 x ULN
* Adequately controlled type 1 or 2 diabetic subjects

Exclusion Criteria:

* Islet cell, acinar cell carcinoma, non-adenocarcinoma (eg, lymphoma, sarcoma, etc), adenocarcinoma originated from biliary tree or cystadenocarcinoma
* Known central nervous system metastases
* Uncontrolled cardiac disease or any other co-morbid disease that would increase the risk of toxicity
* Adjuvant chemotherapy or chemoradiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2007-06; Primary Completion 2010-01 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (40):
- United States (40):
  - Research Site, Alhambra, California
  - Research Site, Bakersfield, California
  - Research Site, Fullerton, California
  - Research Site, La Jolla, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Northridge, California
  - Research Site, Oxnard, California
  - Research Site, Rancho Mirage, California
  - Research Site, Redondo Beach, California
  - Research Site, San Francisco, California
  - Research Site, Santa Maria, California
  - Research Site, Santa Monica, California
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Marietta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Harvey, Illinois
  - Research Site, Baltimore, Maryland
  - Research Site, Westminster, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, Henderson, Nevada
  - Research Site, Albany, New York
  - Research Site, New York, New York
  - Research Site, Durham, North Carolina
  - Research Site, Hickory, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Eugene, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Greenville, South Carolina
  - Research Site, Austin, Texas
  - Research Site, Dallas, Texas
  - Research Site, Round Rock, Texas
  - Research Site, Tyler, Texas
  - Research Site, Tacoma, Washington
  - Research Site, Yakima, Washington

REFERENCES:
- [Background] Cella D, Butt Z, Kindler HL, Fuchs CS, Bray S, Barlev A, Oglesby A. Validity of the FACT Hepatobiliary (FACT-Hep) questionnaire for assessing disease-related symptoms and health-related quality of life in patients with metastatic pancreatic cancer. Qual Life Res. 2013 Jun;22(5):1105-12. doi: 10.1007/s11136-012-0217-4. Epub 2012 Jun 8. PMID 22678353
- [Background] Kindler HL, Richards DA, Garbo LE, Garon EB, Stephenson JJ Jr, Rocha-Lima CM, Safran H, Chan D, Kocs DM, Galimi F, McGreivy J, Bray SL, Hei Y, Feigal EG, Loh E, Fuchs CS. A randomized, placebo-controlled phase 2 study of ganitumab (AMG 479) or conatumumab (AMG 655) in combination with gemcitabine in patients with metastatic pancreatic cancer. Ann Oncol. 2012 Nov;23(11):2834-2842. doi: 10.1093/annonc/mds142. Epub 2012 Jun 13. PMID 22700995
- [Background] Lu, JF.Exposure-response analysis to facilitate phase 3 dose selection for Ganitumumab (AMG 479) in combination with Gemcitabine to treat metastatic pancreatic cancer.Journal-000728;
- [Background] McCaffery I, Tudor Y, Deng H, Tang R, Suzuki S, Badola S, Kindler HL, Fuchs CS, Loh E, Patterson SD, Chen L, Gansert JL. Putative predictive biomarkers of survival in patients with metastatic pancreatic adenocarcinoma treated with gemcitabine and ganitumab, an IGF1R inhibitor. Clin Cancer Res. 2013 Aug 1;19(15):4282-9. doi: 10.1158/1078-0432.CCR-12-1840. Epub 2013 Jun 5. PMID 23741071
- [Background] TBD.Validation of the FACT-hepatobiliary questionnaire in metastatic pancreatic cancer population.Journal-004521;
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phase 1b AMG 655 3mg/kg | Phase 1b AMG 655 10mg/kg | Phase 2 AMG 655 | Phase 2 AMG 479 | Phase 2 AMG 655-placebo
Started | 6 | 7 | 41 | 42 | 42
Completed | 1 | 0 | 4 | 8 | 3
Not Completed | 5 | 7 | 37 | 34 | 39
Not completed — Adverse Event | 0 | 1 | 5 | 4 | 2
Not completed — Disease progression | 5 | 6 | 27 | 22 | 31
Not completed — Never received IP | 0 | 0 | 0 | 2 | 2
Not completed — Ineligibility determined | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 1 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 4 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1b AMG 655 3mg/kg | Phase 1b AMG 655 10mg/kg | Phase 2 AMG 655 | Phase 2 AMG 479 | Phase 2 AMG 655-placebo | Total
Number analyzed (Participants) | 6 | 7 | 41 | 42 | 42 | 138
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Phase 1b and Phase 2 were not analyzed together.
  years
    Phase 1b: number analyzed (Participants) | 6 | 7 | 0 | 0 | 0 | 13
    Phase 1b | 67.2 (10.7) | 63.7 (15.1) |  |  |  | 65.3 (12.8)
    Phase 2: number analyzed (Participants) | 0 | 0 | 41 | 42 | 42 | 125
    Phase 2 |  |  | 62.3 (9.3) | 62.1 (11.5) | 62.6 (9.1) | 62.3 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 17 | 17 | 16 | 58
  Male | 2 | 3 | 24 | 25 | 26 | 80
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 3 | 3 | 3 | 10
  White | 6 | 6 | 32 | 35 | 37 | 116
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 5 | 4 | 2 | 11
Metastatic pancreatic cancer [Count of Participants; unit: Participants] | 6 | 7 | 41 | 42 | 42 | 138

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs; Phase 1b Portion Only)
Description: The incidence of adverse events and clinical laboratory abnormalities defined as DLTs. A DLT was defined as any grade 3 or higher hematologic or non-hematologic toxicity related to any study treatment.
Time Frame: 28 days
Population: The DLT analysis set consisted of subjects in the phase 1b portion of the study only, who experienced at least 1 DLT in the first 28 days of treatment or received 2 doses of AMG 655, 3 infusions of gemcitabine in a 28 day cycle at doses not less than 750 mg/m2 and were followed for at least 28 days (with or without DLTs).
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b AMG 655 3mg/kg | Phase 1b AMG 655 10mg/kg
Number analyzed (Participants) | 6 | 7
Participants | 0 | 0

2. Primary Outcome: Six Month Overall Survival Rate (Phase 2 Portion Only)
Description: The proportion of subjects alive at 6 months
Time Frame: 6 months
Population: Full analysis (The full analysis set consisted of all randomized subjects in the phase 2 portion of the study, with subjects analyzed according to the randomized treatment.)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2 AMG 655 | Phase 2 AMG 479 | Phase 2 AMG 655-placebo
Number analyzed (Participants) | 41 | 42 | 42
percentage of participants | 59.2 [42.3 to 72.7] | 56.6 [40.8 to 69.7] | 49.5 [33.4 to 63.7]

3. Secondary Outcome: Objective Response Rate
Description: Objective response was defined as a tumor response assessment of either complete response or partial response per modified Response Evaluation Criteria in Solid Tumors [RECIST] and was determined only for subjects with measurable disease at baseline. Per RECIST: a complete response is the disappearance of all target lesions; a partial response is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From start of study treatment through up to 36 months
Population: The Safety Analysis Set for Phase 1b (the safety analysis set consisted of all subjects who received at least 1 dose of investigational product, with subjects analyzed according to the treatment received), and the Full Analysis for Phase 2 (the full analysis set consisted of all randomized subjects in the phase 2 portion of the study, with subjects analyzed according to the randomized treatment).
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Phase 1b AMG 655 3mg/kg | Phase 1b AMG 655 10mg/kg | Phase 2 AMG 655 | Phase 2 AMG 479 | Phase 2 AMG 655-placebo
Number analyzed (Participants) | 6 | 7 | 38 | 39 | 40
percentage of responders | 16.67 [0.42 to 64.12] | 14.29 [0.36 to 57.87] | 2.63 [0.07 to 13.81] | 10.26 [2.87 to 24.22] | 2.50 [0.06 to 13.16]

4. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from study day 1 (phase 1b portion) or randomization (phase 2 portion) to the first observation of disease progression per investigator review (as classified by modified RECIST or clinical progression, whichever occurred first) or death due to any cause, or censoring. Disease progression per RECIST is defined as at least a 20% increase in the sum of diameters of target lesions in reference to the smallest sum on study and an absolute increase of at least 5 mm; the appearance of any new lesions is also considered progression.
Time Frame: From start of study treatment through up to 36 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1b AMG 655 3mg/kg | Phase 1b AMG 655 10mg/kg | Phase 2 AMG 655 | Phase 2 AMG 479 | Phase 2 AMG 655-placebo
Number analyzed (Participants) | 6 | 7 | 41 | 42 | 42
Months | 5.4 [5.3 to 5.6] | 3.5 [1.8 to 13.4] | 3.9 [3.4 to 5.4] | 5.1 [3.2 to 6.0] | 2.1 [1.9 to 3.3]

5. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from study day 1 (phase 1b portion) or randomization (phase 2 portion) to death for any cause.
Time Frame: From start of study treatment through up to 36 months
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1b AMG 655 3mg/kg | Phase 1b AMG 655 10mg/kg | Phase 2 AMG 655 | Phase 2 AMG 479 | Phase 2 AMG 655-placebo
Number analyzed (Participants) | 6 | 7 | 41 | 42 | 42
Months | 9.0 [5.6 to 17.0] | 8.9 [6.9 to 18.5] | 7.5 [4.8 to 10.0] | 8.7 [5.3 to 12.2] | 5.9 [4.1 to 9.7]

6. Secondary Outcome: Number of Subjects With an Adverse Event
Description: Graded Using the National Cancer Institute(NCI) Common Terminology Criteria for Adverse Events(CTCAE) Version 3.0
Time Frame: From start of study treatment through up to 44 weeks
Population: The safety analysis set consisted of all subjects who received at least 1 dose of investigational product, with subjects analyzed according to the treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b AMG 655 3mg/kg | Phase 1b AMG 655 10mg/kg | Phase 2 AMG 655 | Phase 2 AMG 479 | Phase 2 AMG 655-placebo
Number analyzed (Participants) | 6 | 7 | 41 | 40 | 40
Participants | 6 | 7 | 41 | 39 | 40

7. Secondary Outcome: Pharmacokinetics of AMG 655, Ganitumab, and Gemcitabine
Description: PK parameter of Cmax for AMG 655 (phase 1b and phase 2 portions) - pg 266, ganitumab (phase 2 portion only) - pg 270 , and gemcitabine (phase 1b portion only - pg 272) PK parameters
Time Frame: From start of study treatment through up to 48 weeks
Population: The pharmacokinetic analysis set consisted of all subjects who underwent blood sampling for pharmacokinetic evaluation during the study. Cmax for AMG 655 was not calculated for the Phase 2 AMG 479 group because they did not receive AMG 655. The CMAX for AMG479 was not calculated for Phase 1b groups or the Phase 2 AMG 655 groups because they did not receive AMG 479. CMAX of gemcitabine for day 1 and day 8 were only performed in Phase 1b per protocol.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Phase 1b AMG 655 3mg/kg | Phase 1b AMG 655 10mg/kg | Phase 2 AMG 655 | Phase 2 AMG 479
Number analyzed (Participants) | 5 | 6 | 11 | 13
μg/mL
  Cmax for AMG 655: number analyzed (Participants) | 5 | 6 | 11 | 0
  Cmax for AMG 655 | 55.3 (11.3) | 198 (32.5) | 198 (52.7) |
  Cmax for AMG 479: number analyzed (Participants) | 0 | 0 | 0 | 13
  Cmax for AMG 479 |  |  |  | 179 (55.2)
  Cmax for gemcitabine - Day 1: number analyzed (Participants) | 5 | 6 | 0 | 0
  Cmax for gemcitabine - Day 1 | 15.7 (7.79) | 14.8 (7.84) |  |
  Cmax for gemcitabine - Day 8: number analyzed (Participants) | 5 | 6 | 0 | 0
  Cmax for gemcitabine - Day 8 | 10.5 (5.90) | 11.2 (5.76) |  |

8. Secondary Outcome: Dose Intensity of Gemcitabine (Phase 2 Portion Only)
Description: Average Dose intensity of gemcitabine when combined with AMG 655, placebo or AMG 479
Time Frame: From start of study treatment through up to 40 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg/m^2 /infusion
Arm/Group | Phase 2 AMG 655 | Phase 2 AMG 479 | Phase 2 AMG 655-placebo
Number analyzed (Participants) | 41 | 40 | 40
mg/m^2 /infusion | 861.40 (119.45) | 906.66 (115.76) | 936.29 (79.58)

9. Secondary Outcome: Duration of Response
Description: Duration of response was the time from the first observation of an objective response to the subsequent time of disease progression (per modified RECIST or clinical progression, whichever came first) or death due to any cause. Objective response = a tumor response assessment of either complete response or partial response per modified Response Evaluation Criteria in Solid Tumors [RECIST]. Per RECIST: a complete response is the disappearance of all target lesions; a partial response is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From objective response through up to 36 months
Population: Only subjects with a CR or PR were analyzed. Duration of response was only measured for Phase 2.
Measure: Median (Full Range); unit: Days
Arm/Group | Phase 1b AMG 655 3mg/kg | Phase 1b AMG 655 10mg/kg | Phase 2 AMG 655 | Phase 2 AMG 479 | Phase 2 AMG 655-placebo
Number analyzed (Participants) | 0 | 0 | 1 | 4 | 1
Days |  |  | 301 [301 to 301] | 253 [60 to 472] | 116 [116 to 116]

10. Secondary Outcome: Incidence of Antibody Formation
Description: The incidence of antibody formation of anti-AMG 655 (phase 1b and phase 2 portions) or anti- ganitumab (phase 2 portion only)
Time Frame: From start of treatment up to 40 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b AMG 655 3mg/kg | Phase 1b AMG 655 10mg/kg | Phase 2 AMG 655 | Phase 2 AMG 479 | Phase 2 AMG 655-placebo
Number analyzed (Participants) | 6 | 7 | 41 | 42 | 42
Participants | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were measured from start of study treatment up to 44 weeks. Mortality was measured from start of treatment to up to 36 months.
Description: The safety analysis set was used for adverse events, which consisted of all subjects who received at least 1 dose of investigational product, with subjects analyzed according to the treatment received. The full population was used for mortality.
Arm/Group | Phase 1b AMG 655 3mg/kg | Phase 1b AMG 655 10mg/kg | Phase 2 AMG 655 | Phase 2 AMG 479 | Phase 2 AMG 655-placebo
All-Cause Mortality (participants affected / at risk) | 5/6 | 7/7 | 32/41 | 28/42 | 33/42
Serious Adverse Events (participants affected / at risk) | 4/6 | 4/7 | 23/41 | 21/40 | 20/40
Other Adverse Events (participants affected / at risk) | 6/6 | 7/7 | 41/41 | 39/40 | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b AMG 655 3mg/kg (N=6) | Phase 1b AMG 655 10mg/kg (N=7) | Phase 2 AMG 655 (N=41) | Phase 2 AMG 479 (N=40) | Phase 2 AMG 655-placebo (N=40)
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 2 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 2 | 3 | 2 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 1 | 0
Infusion Related Reaction (General disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 1 | 4 | 3 | 2
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Bilateral Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 1
Pancreatic Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Mental Status Changes (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 2
Deep Vein Thrombosis (Vascular disorders) | 1 | 1 | 2 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Angina Pectoris (Cardiac disorders) | 0 | 0 | 2 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Optic Ischaemic Neuropathy (Eye disorders) | 0 | 0 | 0 | 0 | 1
Duodenal Obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Gastric Perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Obstruction Gastric (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 0
Death (General disorders) | 0 | 0 | 1 | 0 | 0
Disease Progression (General disorders) | 0 | 0 | 0 | 0 | 2
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1
Generalised Oedema (General disorders) | 0 | 0 | 0 | 1 | 0
Oedema Peripheral (General disorders) | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1 | 0 | 0
Bile Duct Obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1
Hepatic Failure (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 1
Catheter Related Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 2
Clostridium Difficile Colitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Stent Occlusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Blood Bilirubin Increased (Investigations) | 0 | 0 | 0 | 1 | 0
Lipase Increased (Investigations) | 0 | 0 | 1 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Primary Tumor (General disorders) | 0 | 0 | 0 | 1 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Malignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 3
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0
Carotid Artery Stenosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Embolic Stroke (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Hepatic Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Reversible Posterior Leukoencephalopathy Syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Renal Failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 0 | 0 | 1 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 1 | 0
Jugular Vein Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Peripheral Embolism (Vascular disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b AMG 655 3mg/kg (N=6) | Phase 1b AMG 655 10mg/kg (N=7) | Phase 2 AMG 655 (N=41) | Phase 2 AMG 479 (N=40) | Phase 2 AMG 655-placebo (N=40)
Anaemia (Blood and lymphatic system disorders) | 2 | 3 | 12 | 9 | 14
Hypercoagulation (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2 | 2 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 3 | 0 | 13 | 10 | 9
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 3 | 18 | 14 | 14
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 2 | 0 | 0 | 1
Sinus Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Dry Eye (Eye disorders) | 1 | 0 | 0 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2
Abdominal Pain (Gastrointestinal disorders) | 2 | 5 | 8 | 6 | 11
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0 | 4 | 6 | 4
Constipation (Gastrointestinal disorders) | 3 | 4 | 16 | 18 | 18
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 11 | 8 | 6
Dry Mouth (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 3 | 3 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 2 | 2 | 2
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 5 | 14 | 22 | 25
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 4 | 10 | 14 | 9
Asthenia (General disorders) | 0 | 2 | 3 | 5 | 2
Catheter Site Haemorrhage (General disorders) | 0 | 1 | 0 | 0 | 0
Chest Pain (General disorders) | 1 | 1 | 3 | 3 | 1
Chills (General disorders) | 1 | 0 | 5 | 6 | 8
Early Satiety (General disorders) | 1 | 1 | 1 | 0 | 0
Fatigue (General disorders) | 5 | 7 | 26 | 19 | 22
Infusion Related Reaction (General disorders) | 1 | 0 | 0 | 0 | 0
Infusion Site Mass (General disorders) | 1 | 0 | 0 | 0 | 0
Infusion Site Pain (General disorders) | 1 | 0 | 0 | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 1 | 0 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 2 | 2 | 14 | 11 | 10
Pain (General disorders) | 0 | 1 | 4 | 7 | 6
Pyrexia (General disorders) | 3 | 1 | 14 | 8 | 15
Ear Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Otitis Externa (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1 | 1
Sepsis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 1 | 0 | 2 | 2
Urinary Tract Infection (Infections and infestations) | 1 | 2 | 2 | 3 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1 | 0
Joint Dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Skeletal Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Stent Occlusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 2
Ejection Fraction Decreased (Investigations) | 0 | 1 | 0 | 0 | 0
International Normalised Ratio Increased (Investigations) | 0 | 1 | 1 | 0 | 1
Lipase Increased (Investigations) | 0 | 1 | 3 | 0 | 2
Neutrophil Count Increased (Investigations) | 0 | 1 | 1 | 2 | 1
Waist Circumference Increased (Investigations) | 0 | 1 | 0 | 0 | 0
Weight Decreased (Investigations) | 1 | 2 | 3 | 6 | 3
Weight Increased (Investigations) | 0 | 1 | 1 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 3 | 8 | 12 | 13
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 4 | 10 | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 3 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 4 | 5 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 2 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2 | 3 | 2 | 2
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 3 | 1
Bilateral Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4 | 4 | 4
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4 | 0 | 0
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 1 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 0
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 3 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 2 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 6 | 0 | 2
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 1
Pancreatic Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 1
Burning Sensation (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 4 | 4 | 3
Memory Impairment (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 7 | 5 | 6
Blunted Affect (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Depressed Mood (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 2 | 1 | 5 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 5 | 4 | 8
Mental Status Changes (Psychiatric disorders) | 0 | 1 | 1 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1
Bladder Neck Obstruction (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 2 | 0 | 5
Renal Failure (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0
Urinary Hesitation (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Breast Pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 9 | 3 | 11
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 1
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2 | 3
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 3
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 5 | 7 | 3
Rash Papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 1 | 5 | 2 | 1
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hot Flush (Vascular disorders) | 0 | 2 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 2 | 2 | 2
Hypotension (Vascular disorders) | 0 | 3 | 6 | 5 | 4
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 4 | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 3
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Angina Pectoris (Cardiac disorders) | 0 | 0 | 2 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 2 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 1 | 0
Eye Irritation (Eye disorders) | 0 | 0 | 0 | 1 | 0
Ocular Icterus (Eye disorders) | 0 | 0 | 1 | 1 | 0
Optic Ischaemic Neuropathy (Eye disorders) | 0 | 0 | 0 | 0 | 1
Photophobia (Eye disorders) | 0 | 0 | 2 | 0 | 0
Vision Blurred (Eye disorders) | 0 | 0 | 1 | 2 | 1
Visual Impairment (Eye disorders) | 0 | 0 | 0 | 1 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 2 | 5 | 5
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 4 | 2 | 3
Duodenal Obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Epigastric Discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1
Faecal Incontinence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Faeces Discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastric Perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastrointestinal Sounds Abnormal (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 3 | 2 | 4
Gingival Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Hiatus Hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Lip Dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Obstruction Gastric (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Oral Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pancreatic Enzyme Abnormality (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pancreatic Insufficiency (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Sensitivity Of Teeth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 1
Tooth Disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Varices Oesophageal (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Catheter Site Pain (General disorders) | 0 | 0 | 1 | 1 | 0
Chest Discomfort (General disorders) | 0 | 0 | 0 | 1 | 1
Death (General disorders) | 0 | 0 | 1 | 0 | 0
Disease Progression (General disorders) | 0 | 0 | 0 | 0 | 2
Gait Disturbance (General disorders) | 0 | 0 | 1 | 0 | 1
Generalised Oedema (General disorders) | 0 | 0 | 0 | 1 | 0
Hernia (General disorders) | 0 | 0 | 0 | 1 | 0
Influenza Like Illness (General disorders) | 0 | 0 | 1 | 0 | 2
Infusion Site Hypersensitivity (General disorders) | 0 | 0 | 0 | 1 | 0
Injection Site Reaction (General disorders) | 0 | 0 | 1 | 0 | 2
Localised Oedema (General disorders) | 0 | 0 | 0 | 1 | 1
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0
Mucosal Inflammation (General disorders) | 0 | 0 | 3 | 0 | 1
Oedema (General disorders) | 0 | 0 | 2 | 0 | 0
Temperature Intolerance (General disorders) | 0 | 0 | 1 | 0 | 0
Bile Duct Obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1
Hepatic Failure (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 4 | 3 | 3
Jaundice (Hepatobiliary disorders) | 0 | 0 | 2 | 2 | 1
Biliary Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Candidiasis (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Catheter Related Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 2 | 1 | 2
Clostridium Difficile Colitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Herpes Virus Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Infected Cyst (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Localised Infection (Infections and infestations) | 0 | 0 | 2 | 1 | 0
Lung Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Oral Candidiasis (Infections and infestations) | 0 | 0 | 2 | 1 | 0
Oral Herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Postoperative Wound Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 2 | 0 | 1
Viral Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Vulvovaginal Mycotic Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Incision Site Pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Open Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Tooth Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0
Upper Limb Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Alanine Aminotransferase (Investigations) | 0 | 0 | 1 | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 5 | 6 | 7
Aspartate Aminotransferase (Investigations) | 0 | 0 | 1 | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 5 | 6 | 8
Blood Albumin Decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood Alkaline Phosphatase (Investigations) | 0 | 0 | 0 | 1 | 2
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 0 | 1 | 3 | 3
Blood Amylase (Investigations) | 0 | 0 | 1 | 0 | 1
Blood Amylase Increased (Investigations) | 0 | 0 | 3 | 0 | 0
Blood Bilirubin (Investigations) | 0 | 0 | 0 | 0 | 1
Blood Bilirubin Increased (Investigations) | 0 | 0 | 3 | 1 | 2
Blood Calcium Decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood Cholesterol (Investigations) | 0 | 0 | 0 | 0 | 1
Blood Cholesterol Increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood Creatinine (Investigations) | 0 | 0 | 0 | 2 | 0
Blood Glucose Increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood Magnesium Decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood Potassium Increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood Pressure Increased (Investigations) | 0 | 0 | 0 | 1 | 0
Blood Sodium Decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood Uric Acid Increased (Investigations) | 0 | 0 | 1 | 0 | 1
Glomerular Filtration Rate Decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Glucose Urine Present (Investigations) | 0 | 0 | 0 | 1 | 0
Haemoglobin (Investigations) | 0 | 0 | 2 | 0 | 1
Haemoglobin Decreased (Investigations) | 0 | 0 | 3 | 6 | 3
Heart Rate Increased (Investigations) | 0 | 0 | 0 | 1 | 0
Lipase (Investigations) | 0 | 0 | 1 | 0 | 1
Neutrophil Count (Investigations) | 0 | 0 | 1 | 1 | 1
Platelet Count Decreased (Investigations) | 0 | 0 | 2 | 3 | 2
White Blood Cell Count Decreased (Investigations) | 0 | 0 | 3 | 2 | 3
White Blood Cell Count Increased (Investigations) | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 7 | 6 | 5
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Fluid Retention (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 4 | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Primary Tumor (General disorders) | 0 | 0 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscle Fatigue (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Choroid Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Malignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 3
Metastases To Liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
Carotid Artery Stenosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Dementia Alzheimer's Type (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 4 | 3 | 6
Dysgeusia (Nervous system disorders) | 0 | 0 | 5 | 3 | 2
Embolic Stroke (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Hepatic Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 2 | 1 | 0
Neuropathy Peripheral (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Reversible Posterior Leukoencephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 2 | 0
Syncope (Nervous system disorders) | 0 | 0 | 2 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Anxiety Disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Confusional State (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0
Choluria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 2
Hypertonic Bladder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Renal Failure Acute (Renal and urinary disorders) | 0 | 0 | 1 | 2 | 0
Urge Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Amenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Scrotal Oedema (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 4 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 1 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Increased Upper Airway Secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3 | 0
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Cold Sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1
Pain Of Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
Capillary Leak Syndrome (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Jugular Vein Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Orthostatic Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Orthostatic Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Peripheral Embolism (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 2
Phlebitis Superficial (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 1
Vasodilatation (Vascular disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2008-11-20): https://cdn.clinicaltrials.gov/large-docs/52/NCT00630552/Prot_SAP_000.pdf